CLINICAL TRIAL: NCT00177359
Title: Restoring Skill in Walking
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0508137
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2007-12-13 (Estimated); Status verified 2007-12

CONDITIONS: Mobility Limitation
Keywords: gait impairment
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: gait intervention

SUMMARY:
The purpose of the study is to examine the effect of an intervention to improve walking based on motor learning (skill-based) compared to the usual intervention (strength, flexibility and balance-based) on clinical, psychological and laboratory measures of walking and balance of older adults with mobility disability (walking problems).

DETAILED DESCRIPTION:
While therapeutic exercise to improve mobility and balance appears to improve physical performance and may reduce falls, less is known about the responsiveness to specific interventions or the relation between response to intervention and the underlying problems or impairments. Therapeutic approaches for improving mobility and reducing fall risk are heterogeneous, but do not consistently focus on problem solving as a method of enhancing motor control or skill, an approach that has been found to be important for motor learning in animal models.

This two-year pilot study will allows us to compare the clinical, psychological and laboratory outcomes after a motor-learning based and an impairment-targeted exercise intervention to improve walking in older adults. All subjects will participate in pre and post intervention testing and a 12 week exercise intervention for gait involving either a motor learning (skill enhancement) or impairment-targeted (lower extremity strengthening, flexibility and gait cues).

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age and older
* Ambulatory (with or without a straight cane, and without the assistance of another person)
* Have written approval/clearance of their physician to participate in low to moderate intensity, supervised exercise as is characteristic of the interventions for improving gait.
* Difficulty with walking or balance as indicated by the following two criteria during baseline testing:

  * mild to moderate slowing of walking speed (walking speed ≥ .6m/s and ≤ 1.0m/s) and,
  * gait variability (step length coefficient of variability, CV > 4.5%, or step width CV < 7% or > 30%)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2005-11; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Change in gait variability, energy cost of walking, perception of effort in walking, and adaptability of gait to changing environmental conditions, pre and post intervention (12 weeks)

SECONDARY OUTCOMES:
Physical activity, endurance in walking, falls efficacy, performance of usual activities of living, pre and post intervention (12 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Jessie VanSwearingen, PhD, PT, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] VanSwearingen JM, Perera S, Brach JS, Wert D, Studenski SA. Impact of exercise to improve gait efficiency on activity and participation in older adults with mobility limitations: a randomized controlled trial. Phys Ther. 2011 Dec;91(12):1740-51. doi: 10.2522/ptj.20100391. Epub 2011 Oct 14. PMID 22003158